CLINICAL TRIAL: NCT03708081
Title: Comparative Evaluation of Different File Systems in Postoperative Pain: Randomize Clinical Study
Brief Title: Comparative Evaluation of Different File Systems in Postoperative Pain
Status: Completed | Type: Observational
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Mustafa Murat Koçak, Associate professor, Bulent Ecevit University
Other Study IDs: BEU
Record Dates: First submitted 2018-10-11; First posted 2018-10-17 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Pulpitis; Periapical Periodontitis; Necrotic Pulp
MeSH Terms: conditions — Pulpitis; Periapical Periodontitis; Dental Pulp Necrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Root canal treatments will be completed by ProTaper Next instruments with rotational motion
  Interventions: Procedure: ProTaper Next
- Group 2: Root canal treatments will be completed TF Adaptive instruments with adaptive motion.
  Interventions: Procedure: TF Adaptive

INTERVENTIONS:
Procedure: ProTaper Next — Root canal instrument
  Groups: Group 1
Procedure: TF Adaptive — Root canal instrument
  Groups: Group 2

SUMMARY:
Postoperative pain is a frequent complication associated with root canal treatment. The apical extrusion of irrigant and debris, including bacteria and necrotic tissue, may lead to postoperative pain, periapical inflammation, and flare-ups. The instrumentation technique and the file design may affect the amount of debris extrusion.

The aim of this study was to evaluate the influence of instrumentation techniques on the incidence and intensity of postoperative pain after single-visit root canal treatment.

DETAILED DESCRIPTION:
Sixty patients having root canal treatment indication and a single root canal were included in the study. The patients were randomly assigned into 2 groups according to root canal instrumentation technique used. In group 1; ProTaper Next (Dentsply Maillefer, Ballaigues, Switzerland) instruments with rotational motion, in group 2 TF Adaptive (SybronEndo, Orange, CA) instruments with adaptive motion were used for root canal treatments. Root canal treatment was carried out in a single visit and the severity of postoperative pain was assessed via a four-point pain intensity scale. All the participants were called through the phone at 12, 24 and 48h to obtain the pain scores. Data were analyzed using the Mann Whitney-U, Friedman and Wilcoxon tests.

ELIGIBILITY:
Inclusion Criteria:

* having root canal treatment indication
* single root canal

Exclusion Criteria:

* previously treated tooth

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients referred to dental clinic for endodontic treatment
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2018-10-05 (Actual)

PRIMARY OUTCOMES:
Post operative pain | 2 days
  Postoperative pain which occurs after root canal instrumentation and measured with a commonly used scale named 'four-point pain intensity scale' for pain intensity. Patients were instructed postoperatively to express their pain according to the staed scale ranging between no pain and severe pain.
  The scale consists of 4 scores ranging between 1-4. The pain categories were as follows;
  1. no pain;
  2. mild pain (slight discomfort, no need for treatment);
  3. moderate pain (pain relieved by medication);
  4. severe pain (pain and/or swelling not relieved by simple analgesic medication and unscheduled visit required). For patients having no pain score 1, for patients having slight pain in case of no medication score 2 , and score 3 in case of any requirement of medication due to moderate pain, and score 4 for patients having severe pain with the requirement of an unscheduled visit were accepted.
  The higher values represent more pain intensity.

CONTACTS AND LOCATIONS:
Locations (1):
- Bülent Ecevit University, Faculty of Dentistry, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided